CLINICAL TRIAL: NCT00520871
Title: The Effect of Blueberry Juice on Cardiovascular Risk Factors, and Markers of Antioxidant Status, Oxidative Stress Status and Inflammation.
Brief Title: The Water-Blueberry Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Ullevaal University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Water-Blueberry Study; REK SØR ref nr 39-03-01166
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2007-08-27 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Blueberruy; Antioxidants; Oxidative stress; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Blueberry juice

SUMMARY:
We will study the effect of supplementation of 1 L blueberry juice to participants with at least one elevated cardiovasculat risk factor.

DETAILED DESCRIPTION:
Participants with at leat one elevated cardiovacsular risk factor, as defined as systolic blood pressure between 140 and 165 mmHg, diastolic blood pressure between 90 and 105 mmHg, low density lipoprotein (LDL) cholesterol ≥3.4 mmol/L, total/high density lipoprotein (HDL) cholesterol ratio >4 or smoking a minimum of 3 cigarettes daily.

Subjects were randomized to two groups, where the blueberry group were supplemented with 1 L blueberry juice per day for four weeks. The control group consumed an equal amount of water.

Clinical markers, as well as biomarkers of antioxidant status, oxidative stress status and inflammation were measured in blood samples before amd after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years for men and 45-70 years or at least 12 months postmenopausal for women
* at least one elevated cardiovascular risk factor, defined as systolic blood pressure between 140 and 165 mmHg, diastolic blood pressure between 90 and 105 mmHg, low density lipoprotein (LDL) cholesterol ≥3.4 mmol/L, total/high density lipoprotein (HDL) cholesterol ratio >4 or smoking a minimum of 3 cigarettes daily.

Exclusion Criteria:

* clinically recognized chronic diseases as impaired renal function, diabetes mellitus, cardiovascular disease, liver or gastrointestinal disease or cancer within the last 5 years
* use of lipid-lowering drugs, diuretics or hormone replacement therapy for women
* Subjects with a body-mass index ≥31
* with a alcohol consumption above 3 units/day for men and 1 unit/day for women
* blood donation within the last six months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-03; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoints are cardiovascular risk factors | 4 weeks

SECONDARY OUTCOMES:
Secondary endpoints are additional clinical markers, as well as biomarkers of antioxidant status, oxidative stress status and inflammation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rune Blomhoff, PhD, Principal Investigator — University of Oslo; Serena Tonstad, MD, Principal Investigator — Ullevaal University Hospital; Anette Karlsen, MSc, Principal Investigator — University of Oslo